CLINICAL TRIAL: NCT00331786
Title: Phase I Multiple-Dose Safety, Pharmacokinetic and Pharmacodynamic Clinical Study of Nitric Oxide Releasing Aspirin (NCX 4016)
Brief Title: Nitric Oxide-Releasing Acetylsalicyclic Acid in Preventing Colorectal Cancer in Patients at High Risk of Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000473094; SUNY-UH-20055574
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-05

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — nitroaspirin; Biopsy

INTERVENTIONS:
Drug: nitric oxide-releasing acetylsalicylic acid derivative
Other: laboratory biomarker analysis
Procedure: biopsy

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of nitric oxide-releasing acetylsalicyclic acid may prevent colorectal cancer.

PURPOSE: This randomized phase I trial is studying the side effects and best dose of nitric oxide-releasing acetylsalicyclic acid in preventing colorectal cancer in patients at high risk of colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the effects of nitric oxide-releasing acetylsalicyclic acid on aberrant cryptic foci (ACF) in patients at high risk for colon cancer.

Secondary

* Determine the pharmacokinetic profile of this drug in these patients.
* Determine the presence or absence of ACF in these patients.
* Determine the expression of PGE2, COX-1, COX-2, NF-kB, and β-catenin in colon tissue.
* Determine the safety and tolerability of long-term nitric oxide-releasing acetylsalicyclic acid in these patients.

OUTLINE: This is a multicenter, double-blind, randomized, placebo-controlled, parallel group study. Patients are stratified according to gender and race (black vs non-Hispanic white vs Hispanic white vs Asian). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive oral nitric oxide-releasing acetylsalicyclic acid twice daily for 6 months.
* Arm II: Patients receive nitric oxide-releasing acetylsalicyclic acid twice daily for 6 months at a higher dose than in arm I.
* Arm III: Patients receive oral placebo twice daily for 6 months. Patients undergo sigmoidoscopies at baseline and at the completion of study treatment. Biopsies of aberrant cryptic foci (ACF) and non-ACF sites are collected at both sigmoidoscopies. Tissue is examined for biomarkers (PGE_2, COX, NF-kB, β-catenin).

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 240 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At risk for colorectal cancer

  * History of histologically proven sporadic colon adenomas or colon cancer
  * At least 5 aberrant cryptic foci on sigmoidoscopy
  * Less than 20 prior cumulative adenomas and no heredity nonpolyposis colorectal cancer
* No significant asymptomatic lesions on sigmoidoscopy, including any of the following:

  * Inflammation
  * Strictures
  * Anorectal lesions
  * Fistulae
  * Vascular lesions
* No adenomas or colon carcinomas on flexible sigmoidoscopy
* No history of gastrointestinal (GI) cancer other than colorectal cancer
* No inherited colorectal cancer syndromes

PATIENT CHARACTERISTICS:

* No other GI mucosal epithelial diseases (e.g., Barrett's esophagus, chronic or recurrent peptic ulcer disease, celiac sprue, or other disorders of nutrient absorption)

  * No active peptic ulcer disease
* No history of inflammatory bowel disease (ulcerative colitis or Crohn's disease)
* No known or suspected alcohol ( > 5 glasses of wine or beer per day), drug, or medication abuse
* No quantitative or qualitative platelet or coagulation abnormalities
* No personal or family history of a bleeding disorder
* No uncontrolled diabetes
* No uncontrolled hypertension, or chronic congestive heart failure (New York Heart Association class II-IV heart disease)
* No myocardial infarction, transient ischemic attack, or stroke within the past 6 months
* No equilibrium disorders affecting gait or ability to stand that would preclude study participation
* No involuntary change in weight (up or down) of ≥ 15% of usual body weight within the past year
* Creatinine ≤ 2.0 mg/dL
* No chronic liver disease or pancreatitis
* No allergies to aspirin
* No prior severe adverse reactions to NSAIDs such as asthma, GI bleeding, or renal insufficiency
* No institutionalized, mentally disabled patients
* No prisoners
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* No concurrent antibiotic prophylaxis
* More than 7 days since prior nonsteroidal anti-inflammatory drug (NSAID) treatment, including aspirin
* No concurrent frequent use (> 7 days in previous month) of NSAIDs, cyclooxygenase (COX)-2 inhibitors, nitrovasodilators, or oral corticosteroids
* No concurrent macronutrient consumption below the 1st or above the 99th percentile of U.S. consumption
* No concurrent anticoagulants, ticlopidine, and clopidogrel
* More than 3 months since prior general anesthesia
* More than 3 months since prior investigational agents
* No concurrent NSAIDs, including aspirin or COX-2 inhibitors

  * Acetaminophen allowed
* No concurrent nitrovasodilating drugs
* More than 3 months since prior participation in other investigational trials

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2006-07

PRIMARY OUTCOMES:
Effects of nitric oxide-releasing acetylsalicyclic acid (NCX 4016) on aberrant cryptic foci (ACF) multiplicity after the second dose at 6 months

SECONDARY OUTCOMES:
Pharmacokinetic profile by blood, urine, and colon tissue sampling
Incidence of ACF as measured by magnification chromoendoscopy
Assessment of biomarkers expressed in colon tissue, including PGE2 (measured by immunoassay), COX-1, COX-2, NF-kB, and β-catenin (measured by immunohistochemistry) at baseline and at the final visit
Data on C-Reactive protein as a marker for inflammation
Safety and tolerability of long-term oral administration of NCX 4016 as measured by NCI CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Basil Rigas, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Cancer Center, Stony Brook, New York, United States